CLINICAL TRIAL: NCT00935753
Title: Trial of Kuvan™ (Sapropterin) Treatment in Patients With Lesch Nyhan Disease
Brief Title: Trial of Kuvan in Lesch-Nyhan Disease
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Contractual issues
Sponsor: University of California, San Diego (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WLN01
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Behavioral Manifestations of Lesch-Nyhan Disease
Keywords: Lesch-Nyhan Disease; self-mutilating behavior
MeSH Terms: conditions — Lesch-Nyhan Syndrome; Self-Injurious Behavior | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kuvan (Experimental): 10mg/kg Kuvan for 5 days followed by 20mg/kg Kuvan for a total of 60 days
  Interventions: Drug: sapropterin

INTERVENTIONS:
Drug: sapropterin — oral 100mg tablets taken intact or dissolved in water or apple juice with morning meal for up to 60 days

SUMMARY:
To assess the possibility that treatment with Kuvan (a form of tetrahydrobiopterin) will lessen the abnormal behavior and/or neurology commonly found in Lesch-Nyhan disease (LND); to assess biochemical changes as measured in blood and urine.

DETAILED DESCRIPTION:
Lesch-Nyhan disease (LND) is an X-linked disorder of purine metabolism which results from mutation in the gene for the enzyme hypoxanthineguanine phosphoribosyltransferase (HPRT); patients have hyperuricemia, gout, urinary tract calculi, and nephropathy which are effectively treated with allopurinol. There is also a syndrome of dystonia, chorea and athetosis, as well as involuntary self mutilative biting and aggression toward their caretakers, for which there is no treatment.

Kuvan™ is a form of tetrahydrobiopterin (BH4), and is approved to help lower the blood levels of phenylalanine in people who have phenylketonuria (PKU). LND patients have been found to have decreased BH4 in the spinal fluid and brain; BH4 is a precursor of dopamine, which has an effect on behavior. In an earlier study Dr Nyhan found that treatment of LND with 5-hydroxytryptophan and carbidopa abolished the self-injurious behavior but was uniformly transient.

This is a single site open-label protocol for eight subjects age 4 years and older with Lesch-Nyhan Disease documented by deficiency of HPRT.

The study involves three study visits to San Diego and one study visit done locally. The first visit will last 13 days, the following visits are single day visits at week 4 and week 8, and the local study visit is a brief outpatient visit at week 6. Physical and neurological exams, videotaping of the patient's interactions with the study staff, and blood and urine collection for laboratory analyses will be performed at each San Diego visit. A family member or caregiver will be asked to complete a short assessment form and report any illness or medication changes. In addition, the study staff will have weekly telephone contact with the family to discuss any behavioral changes or study drug issues.

If the patient's self injurious behavior becomes worse after starting Kuvan the drug will be discontinued and the patient will be followed until the behavior returns to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 4 years and older
2. Must have documented evidence of HPRT deficiency.
3. Be on a stable treatment regimen for 30 days or more
4. Willing and able to travel to San Diego for the study visits
5. Have a local neurologist or physician familiar with the patient or experienced in managing behavioral/neuromuscular disorders and willing to assist with study procedures and adverse events if necessary

Exclusion Criteria:

1. Concurrent enrollment in an investigational drug study
2. Currently taking levodopa
3. Elevated liver enzymes
4. Renal or liver impairment or disease
5. Inability to comply with required study procedures

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Clinical responses to be monitored will include frequency and severity of self mutilation episodes, frequency and severity of aggressive acts towards others, and any effect on involuntary movements. | Periodically during the eight weeks of treatment per patient

SECONDARY OUTCOMES:
Effect of Kuvan on standard chemistries, plasma amino acids, and plasma and urinary catecholamines | Assessed periodically during treatment

CONTACTS AND LOCATIONS:
Overall Officials: William L Nyhan, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Mitochondrial and Metabolic Disease Center, San Diego, California, United States